CLINICAL TRIAL: NCT04253028
Title: Use of NERv's Inline Device for the Continuous Monitoring of pH and Conductance Measurements as an Early Diagnostic Method for Anastomotic Leak.
Brief Title: Use of NERv's Inline Device as an Early Diagnostic Method for Anastomotic Leak.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: FluidAI Medical (Industry)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLS0005
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Anastomotic Leak
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with NERv's Inline Device Attached (Experimental): This arm contains subjects which will have NERv's Inline Device attached to their peritoneal drain after bariatric surgery (this includes: Roux-en-Y Gastric Bypass (RYGBP), Sleeve Gastrectomy (SG), Gastric Plication and Duodenal Switch).
  Interventions: Device: NERv's Inline Device

INTERVENTIONS:
Device: NERv's Inline Device — NERv's Inline Device attaches to existing catheters or peritoneal drains that are currently being used in the medical industry. This allows the device to measure the pH and conductance of intraperitoneal fluids that typically get drained through peritoneal drains.

SUMMARY:
NERv's early feasibility clinical trial is a first-in-human, multi-center, pre-market, non-randomized clinical trial intended to evaluate the safety and collect preliminary data necessary for the detection of clinical post-operative anastomotic/intraperitoneal leakages.

NERv's Inline Device attaches to existing catheters or peritoneal drains that are currently being used in the medical industry. This allows the device to measure the pH and conductance of intraperitoneal fluids that typically get drained through peritoneal drains.

The purpose of NERv's feasibility clinical trial is to collect pH and conductance readings by analyzing peritoneal drainage fluid. Upon analyzing data collected from NERv's Inline Device a clinical model of pH and conductance will be created. The clinical model can then be used to determine if a complication is developing. For instance, boundaries (reading thresholds) can be established where if the signal goes outside the boundaries a complication could be identified. Specifically the ability to detect a post-operative complication known as anastomotic leakage; which is a dreaded complication associated with abdominal surgeries; will be the main focus of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years - male or female
* Subject understands and has voluntarily signed and dated Informed Consent Form (ICF)
* Subjects must be willing to comply with trial requirements
* Subject has a peritoneal drain attached post-surgery

Exclusion Criteria:

* Plans that the subject will be discharged less than 8 hours post-surgery
* Involvement in the planning and conduct of the clinical investigation
* Subject is participating in another investigational drug or device study which would interfere with the endpoints and follow-ups of this study
* Subject is consuming steroid or anti-inflammatory medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in pH of Peritoneal Fluid | A clinical model of change in pH over time will be established once the study is completed (up to 28 weeks).
  NERv's Inline Device will be collecting continuous pH measurements of fluid that travels across the peritoneal drain of bariatric surgery patients.
Change in Conductance of Peritoneal Fluid | A clinical model of change in conductance over time will be established once the study is completed (up to 28 weeks).
  NERv's Inline Device will be collecting continuous conductance measurements of fluid that travels across the peritoneal drain of bariatric surgery patients.
Change in Temperature of Peritoneal Fluid | A clinical model of change in temperature over time will be established once the study is completed (up to 28 weeks).
  NERv's Inline Device will be collecting continuous temperature measurements of fluid that travels across the peritoneal drain of bariatric surgery patients.
Number of Subjects with Device Related Adverse Events | The number of device related will be established once the study is completed (up to 28 weeks).
  an adverse event assesmtent will be performed in accordance to ISO 14155 standards to determine the number of device related adverse events.

SECONDARY OUTCOMES:
Investigator and Subject Feedback on Device's Ease of Use and Comfort level | Overall comfort level and ease of use will be established once the study is completed (up to 28 weeks).
  Ease of use and comfort levels will be evaluated by collecting responses to a questionnaire that will be filled out by both the investigator/nurse and the subject.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut University Hospital, Cairo
  - Dr. Yosri Gohar Hospital, Cairo